CLINICAL TRIAL: NCT06347757
Title: A 3-Arm Study Comparing the Efficacy of Anti-Reflux Alimentary Reconstruction Protocols (Single-Tract Jejunal Interposition vs Double Tract vs Tube-Like Stomach Reconstruction) After Laparoscopic Proximal Gastrectomy
Brief Title: A 3-Arm Study Comparing the Efficacy of Anti-Reflux Reconstruction Protocols After Laparoscopic Proximal Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, M.D., Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NorthernJiangsuhospital1
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-03

CONDITIONS: Anti-Reflux Alimentary Reconstruction; Laparoscopic Proximal Gastrectomy; Siewert Type II/III Adenocarcinoma of the Esophagogastric Junction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- laparoscopic proximal gastrectomy with single-tract jejunal interposition reconstruction (Experimental)
  Interventions: Procedure: Anti-Reflux Alimentary Reconstruction After Laparoscopic Proximal Gastrectomy
- laparoscopic proximal gastrectomy with double-tract reconstruction (Active Comparator)
  Interventions: Procedure: Anti-Reflux Alimentary Reconstruction After Laparoscopic Proximal Gastrectomy
- laparoscopic proximal gastrectomy with tube-like stomach reconstruction (Active Comparator)
  Interventions: Procedure: Anti-Reflux Alimentary Reconstruction After Laparoscopic Proximal Gastrectomy

INTERVENTIONS:
Procedure: Anti-Reflux Alimentary Reconstruction After Laparoscopic Proximal Gastrectomy — laparoscopic proximal gastrectomy with single-tract jejunal interposition (LPG-STJI) versus double-tract reconstruction (LPG-DTR) versus tube-like stomach reconstruction (LPG-TLR).

SUMMARY:
The efficacy of three different alimentary reconstruction methods after proximal gastrectomy will be investigated in this study in a prospective, multicenter, randomized controlled trial.

DETAILED DESCRIPTION:
In the trial, 180 patients with early upper-third early gastric cancer and Siewert type II/III esophagogastric junction cancer will be enrolled and then randomly assigned to one of three groups: Group A (single-tract jejunal interposition n = 60), Group B (double-tract reconstruction, n = 60), or Group C (tube-like stomach reconstruction, n = 60). The primary co-end points were the incidence of reflux esophagitis at 2 years postoperatively. The secondary end points included the incidence of anastomotic leakage and anastomotic stenosis, operative time, intraoperative blood loss, quality of life, overall survival, and disease-free survival. Quality of life outcomes were assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) 30-item core questionnaire (C30) and the EORTC QLQ stomach cancer-specific questionnaire at 3 months, 12 months, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years old, male or female;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 (indicating fully active and able to continue all predisease activities without restriction) or 1 (indicating restricted in physically strenuous activities but ambulatory and able to perform work of a light or sedentary nature);
3. American Society of Anesthesiology physical status classification of I (indicating normal and healthy), II (indicating mild systemic disease), or III (indicating severe systemic disease);
4. Pathological diagnosis of preoperative endoscopic biopsy: the tumor is located in the upper 1/3 of the stomach (including the esophagogastric junction), and the clinical staging of gastric cancer Ia and Ib (T1N0M0, T1N1M0, and T2N0M0) (14) according to the eighth edition of the AJCC;
5. Patients without contraindications to surgery;
6. Voluntary participation by signing the written informed consent form approved by the institutional review board before study participation;

Exclusion Criteria:

1. Receipt of chemotherapy or radiotherapy for the treatment of GC before either surgical procedure
2. Combined resection required due to other diseases (except cholecystectomy).
3. History of cancer or concurrent cancer in other organs.
4. Previous or current receipt of treatment for systemic inflammatory disease or history of gastrectomy.
5. Patients with coagulation dysfunction which could not be corrected;
6. Vulnerable status (eg, lacking decision-making capacity, pregnant, or planning to become pregnant).
7. Receipt of chemotherapy or radiotherapy before either surgical procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of reflux esophagitis | At 1 year after LPG

SECONDARY OUTCOMES:
Incidence of anastomotic leakage | At 1 year after LPG
Incidence of anastomotic stenosis | At 1 year after LPG
Operative time | Intraoperative
Intra-operative blood loss | Intraoperative
Overall survival, and disease-free survival | At 1 and 3 years after LPG

CONTACTS AND LOCATIONS:
Locations (1):
- Jiajie Zhou, Yangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian Z, Cheng Y, Wang Y, Ren J, Wang S, Wang D. A 3-Arm case-matched analysis of anti-reflux reconstruction methods after laparoscopic proximal gastrectomy - Single tract jejunal interposition vs double tract reconstruction vs tube-like stomach reconstruction. Eur J Surg Oncol. 2025 Feb;51(2):109482. doi: 10.1016/j.ejso.2024.109482. Epub 2024 Nov 19. PMID 39580964